CLINICAL TRIAL: NCT02684968
Title: The Effects of Continuous Bilateral Quadratus Lumborum Analgesia on Pain, Opioid Consumption, and Opioid-related Complications After Open Abdominal Surgery: A Randomized Controlled Trial
Brief Title: Effects of Continuous Bilateral QL Analgesia After Open Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-1273
Record Dates: First submitted 2016-02-11; First posted 2016-02-18 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: local anesthetic continuous infusion (QL block + IV PCA group) or normal saline continuous infusion (IV PCA group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colorectal Surgery with QL block having anesthetic (Experimental): Bilateral QL catheter with local anesthetic infusion + intravenous patient controlled narcotic medication
  Interventions: Procedure: Colorectal surgery
- Colorectal Surgery with QL block having saline (Placebo Comparator): Bilateral QL catheter with normal saline infusion + intravenous patient controlled narcotic medication
  Interventions: Procedure: Colorectal surgery

INTERVENTIONS:
Procedure: Colorectal surgery

SUMMARY:
Eligible patients will be randomized 1:1 without stratification to bilateral continuous QL catheters with local anesthetic continuous infusion (QL block + IV patient-controlled analgesia group) or normal saline continuous infusion (IV patient-controlled analgesia group).

In the postanesthesia care unit (PACU), patients will be given intravenous boluses of hydromorphone or fentanyl as needed. Following immediate recovery from anesthesia, patients will be provided with a hydromorphone IV patient-controlled analgesia pump with standard initial settings and an option of clinician dose for breakthrough pain. IV patient-controlled hydromorphone pump settings will be titrated to comfort level (pain score<4) by blinded clinicians.

Each of the catheters will be connected to patient controlled infusion pump running at a basal rate of 6mL/hour of 0.1% Bupivacaine or normal saline with on-demand bolus of 5 mL every 60 minutes to be started in the operating room before the surgical incision.

Opioid consumption first 72 hours or until discharge, whichever comes first will be recorded.

Pain scores during first 72 hours or until discharge, whichever comes first will be recorded with a verbal rating scale and obtained from the patient's electronic medical records.

The morning of post operative day 1 and post operative day 3 the ORSDS and QOR surveys will be completed.

Morning of the day of discharge, the overall patient satisfaction with pain management survey will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Adults scheduled for elective colorectal surgery with a midline incision;
* American Society of Anesthesiologists (ASA) physical status 1-3.

Exclusion Criteria:

* Contraindication or intolerance to opioids and/or local anesthetics;
* Inability to use IV PCA system;
* History of chronic pain defined as use of opioids for more than 30 consecutive days within the 3 preoperative months at the dose equal or greater than equivalent of 15 mg of morphine and/or abdominal pain for more than 6 months, present most days of the weeks;
* History of neurological illness and/or neuropathy - Peripheral neuropathy, paralysis;
* Pregnancy and/or breastfeeding;
* Chronic renal failure, defined by estimated GFR <60 ml/min;
* Chronic liver failure, defined by cirrhosis, portal hypertension, or history of variceal bleeding.
* BMI > 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Pain Score | The first postoperative pain score with 72 hours or until discharged using the VRS (0-10) scale
  primary hypothesis is that bilateral continuous QL local anesthetic infusion with IV PCA reduces total opioid consumption and/or time-weighted average pain scores during 72 hours after surgery compared to patients under IV PCA alone, and not worse on either outcome. In other words, IV PCA + QL block is superior to IV PCA alone, resulting in lower opioid consumption and/or less pain and not worse on either outcome.
Opioid Consumption | 72 hours after surgery
  primary hypothesis is that bilateral continuous QL local anesthetic infusion with IV PCA reduces total opioid consumption and/or time-weighted average pain scores during 72 hours after surgery compared to patients under IV PCA alone, and not worse on either outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wael Ali Sakr Esa, M.D., Principal Investigator — General Anesthesiology
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No